CLINICAL TRIAL: NCT05196854
Title: Feasibility and Comparison Study of Home Blood Pressure Monitoring and Clinical Hypnosis in Children With Neurofibromatosis Type 1
Brief Title: Clinical Hypnosis and Home Blood Pressure Monitoring in Children With Neurofibromatosis Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 73244
Record Dates: First submitted 2021-12-21; First posted 2022-01-19 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Hypertension; Neurofibromatosis 1; Blood Pressure
Keywords: Procedural Anxiety; Clinical Hypnosis; Neurofibromatosis; Hypertension; Blood pressure monitoring
MeSH Terms: conditions — Hypertension; Neurofibromatosis 1; Neurofibromatoses

STUDY DESIGN:
Intervention Model Description: Randomised Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Standard Blood Pressure measurement at home (Other): Standard home blood pressure measurement at home
  Interventions: Other: Group 1. Standard Home Blood Pressure Measurement
- Group 2. Hypnosis script prior to Home Blood Pressure measurement (Experimental): Participant listens to a pre-recorded hypnosis script (approx 5 mins long) prior to standard home blood pressure measurement.
  Interventions: Other: Group 2. Hypnosis script prior to home blood pressure measurement

INTERVENTIONS:
Other: Group 1. Standard Home Blood Pressure Measurement — Measurement of Blood Pressure using Home blood pressure monitor
  Arms: Group 1: Standard Blood Pressure measurement at home
Other: Group 2. Hypnosis script prior to home blood pressure measurement — Pre-recorded clinical hypnosis script (approx 5 mins long) used prior to standard home blood pressure measurement. Clinical Hypnosis is used as a non-pharmacological technique for reducing procedural anxiety, distress and discomfort with patients.
  Arms: Group 2. Hypnosis script prior to Home Blood Pressure measurement

SUMMARY:
This study has two primary objectives. The first is to determine if it is feasible and reliable for children and families with a diagnosis of Neurofibromatosis Type 1 (NF1) to use of blood pressure (BP) monitor at home.

The second is to determine if there is a difference between a child's measured home BP using standard instructions or using a clinical hypnosis script. This will be determined by a randomised control trial design.

Standard and hypnosis Home BP will be compared to the gold standard measurement of BP measured by a trained health care professional in clinic.

Children who participate will complete a clinic-based BP with a health care professional, then will be randomised into either the standard home BP measurement or using a hypnosis script prior to BP measurement.

DETAILED DESCRIPTION:
Neurofibromatosis Type 1 (NF1) is a rare autosomal dominate genetic disorder that affects an estimated that 1 in 2500 people or 10000 Australians. NF1 affects multiple systems throughout the body. The prevalence of hypertension(HTN) in children and adolescents in the general population is approximately 3.5%. Children and adolescents with a diagnosis of NF1 have an increased incidence of HTN, and has been documented as high as 6.1% to 12%. This is two times higher than the general population.

Clinical adherence to the recommendation of recording annual blood pressure on patients has not been audited. The anecdotal experience of the authors is that most children do not have annual blood pressure (BP) measurements. With the increased uptake of telehealth following the COVID-19 pandemic, children and families may not be reviewed in person for significant periods of time as they prefer consultations over telehealth. As a result, children may miss having their annual blood pressure measured. As a young people with a diagnosis of NF1 have twice the risk of HTN, annual BP measurement is essential.

The American Academy Paediatrics guideline outlines the best practice for BP measurement to ensure true BP reading: The child should be seated in a quiet room for 3-5 minutes before measurement, with back supported and feet uncrossed on the floor. The blood pressure should be measured on the right arm, using the correct sized cuff. This should be completed by a trained clinician. As part of this study, all participants will have a manual sphygmomanometer in clinic-based BP taken on day of recruitment.

One of the primary objectives of this study is to determine if is feasible to use home blood pressure monitoring to screen children with NF1 for hypertension.

Clinical Hypnosis is used as a non-pharmacological technique for reducing procedural anxiety, distress and discomfort with patients. Hypnosis scripts have been successfully used as non-pharmacological adjuncts to reduce pain and anxiety in adult patients undergoing interventional radiological procedures, demonstrating that the benefits of hypnosis techniques can be accessible to patients with little or no training or preparation. Furthermore, healthcare workers who are not experts in hypnosis can be trained to deliver scripts effectively.

If a hypnosis script used while taking home blood pressure readings allows for a calm child and an equivalent clinic BP measure, hypnosis script and home BP monitoring could have greater application across the Royal Children's Hospital.

Therefore the second aim of the study is to see if there is a difference in a child's BP measurements comparing a standard home BP measurement or utilising a calming hypnosis script prior to home BP measurement. This will be compared to the gold standard clinic-based BP measurement completed by a trained professional. The child's self-reported level of anxiety using the Children's Anxiety Meter Scale (CAM-S) will be measured after every BP measurement. In addition, family's perceptions of the process of home BP monitoring will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Is between the ages of 5 and 18 years old at enrolment.
* Has a diagnosis of neurofibromatosis type 1(NF1), confirmed by a physician, and usually attends the NF clinic at The Royal Children's Hospital, Melbourne, Australia (RCH). Including children with known kidney and cardiac disease.
* Primary residence and residential postal address in Victoria.
* The child can sit quietly for 10-15 minutes at home to complete a blood pressure assessment.
* Provide a signed and dated participant and/or parent guardian information and consent form and or has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf.
* For inclusive diverse study group, Parent/caregiver who require an interpreter can be enrolled in this study. Only inhouse interpreter services able to be included,

Exclusion Criteria:

* Has clinically significant cognitive impairment or attention disorder preventing ability to sit in a chair for 15 minutes
* Has confirmed hypertension on previous testing
* Parent/caregiver who require an interpreter and cannot upload BP and Heart rate (HR) values online independently will be excluded from the study.
* Parent/caregiver requiring an interpreter, but the interpreter not present within the face-to-face appointment eg, phone interpreter services.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Day 1. Clinic-based manual sphygmomanometer blood pressure measurement | Day 1. Day of recruitment at the clinic appointment
  Three measures of Systolic/diastolic reading (mmHg) using manual sphygmomanometer by trained professional. Following The American Academy Pediatrics guidelines for best practice for blood pressure (BP) measurement to ensure true BP reading.
Day 1. Clinic-based automatic oscillometer blood pressure measurement | Day 1. Day of recruitment at the clinic appointment
  One reading of systolic/diastolic reading (mmHg) using automatic oscillometer BP monitor by trained professional - Following The American Academy Pediatrics guidelines for best practice for blood pressure (BP) measurement to ensure true BP reading.
Day 2 Home automatic oscillometer blood pressure measurement | Day 2 at home
  Daily measurement of systolic/diastolic (mmHg) home blood pressure(BP) reading (once only) using an automatic home oscillometer BP monitor measurement.
Day 3 Home automatic oscillometer blood pressure measurement | Day 3 at home
  Daily measurement of systolic/diastolic (mmHg) home blood pressure(BP) reading (once only) using an automatic home oscillometer BP monitor measurement.
Day 4 Home automatic oscillometer blood pressure measurement | Day 4 at home
  Daily measurement of systolic/diastolic (mmHg) home blood pressure(BP) reading (once only) using an automatic home oscillometer BP monitor measurement.

SECONDARY OUTCOMES:
Day 1. Clinic-based Children's Anxiety Meter Scale (CAM-S) | Day1 in clinic
  Measurement of participant's reported state of anxiety in clinic when completing BP measurement using Children's Anxiety Meter Scale (CAM-S).
  CAM-S is a state of anxiety patient reported measure. It is coded 0-10 across a vertical analogue scale.
  0 = calm, not nervous or worried 10 = very very nervous and worried
Day 2,3 and 4 Daily Children's Anxiety Meter Scale (CAM-S) score | Daily on Day 2, 3 and 4 at home.
  Daily measure of the participants reported state of anxiety when completing BP measurement at home using Children's Anxiety Meter Scale (CAM-S).
  CAM-S is a state of anxiety patient reported measure. It is coded 0-10 across a vertical analogue scale.
  0 = calm, not nervous or worried 10 = very very nervous and worried
Day 2 Children's Anxiety Meter Scale (CAM-S) score | Day 2 at home.
  Daily measure of the participants reported state of anxiety when completing BP measurement at home using Children's Anxiety Meter Scale (CAM-S).
  CAM-S is a state of anxiety patient reported measure. It is coded 0-10 across a vertical analogue scale.
  0 = calm, not nervous or worried 10 = very very nervous and worried
Day 3 Daily Children's Anxiety Meter Scale (CAM-S) score | Day 3 at home.
  Daily measure of the participants reported state of anxiety when completing BP measurement at home using Children's Anxiety Meter Scale (CAM-S).
  CAM-S is a state of anxiety patient reported measure. It is coded 0-10 across a vertical analogue scale.
  0 = calm, not nervous or worried 10 = very very nervous and worried
Day 4 Children's Anxiety Meter Scale (CAM-S) score | Day 4 at home.
  Daily measure of the participants reported state of anxiety when completing BP measurement at home using Children's Anxiety Meter Scale (CAM-S).
  CAM-S is a state of anxiety patient reported measure. It is coded 0-10 across a vertical analogue scale.
  0 = calm, not nervous or worried 10 = very very nervous and worried
Day 4, Study specific survey of parents/caregivers perceptions | Day 4 only
  Study specific survey. Likert scales used to assess parent/caregiver perception with ease of use of home BP monitor, timeliness to complete measures and interference with family life compared to attending hospital appointment, ease of receiving and returning equipment, and financial cost to attend hospital appointment.
  Data will be reported for each item individually, as the proportion of parents/caregivers who responded positively on the Likert scale, where higher scores indicate less favorable responses.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Dabscheck, MBBS FRACP, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Murdoch Children's Research Institute, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this study will be available six months after publication of the primary outcome.
  The study protocol, analysis plan and consent forms will also be available. The data may obtained from the Murdoch children's Research institute by emailing gabriel.dabscheck@rch.org.au Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the trial steering committee must see and approve the analysis plane describing how the data will be analysed, there must be and agreement around appropriate acknowledgement and and additional costs involve must be covered. Should the trial steering committee be unavailable, this role is delegated to the Murdoch children's Research Institute. Data will only be shared with a recognised research institution which has approved the proposed analysis plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication of primary outcome
Access Criteria: 1. Data access agreement
  2. Approval by Trial Steering Committee
  3. Recognised Research Institute

REFERENCES:
- [Background] Mackay JR, Glenning JP, Grantham BM, Clark K, Mynard JP, Olweny CN, Quinlan C, Dabscheck G. Feasibility of home blood pressure screening in the paediatric outpatient clinic setting. Arch Dis Child. 2025 Jun 19;110(7):551-555. doi: 10.1136/archdischild-2024-327391. PMID 39814532
- [Background] Flynn JT, Kaelber DC, Baker-Smith CM, Blowey D, Carroll AE, Daniels SR, de Ferranti SD, Dionne JM, Falkner B, Flinn SK, Gidding SS, Goodwin C, Leu MG, Powers ME, Rea C, Samuels J, Simasek M, Thaker VV, Urbina EM; SUBCOMMITTEE ON SCREENING AND MANAGEMENT OF HIGH BLOOD PRESSURE IN CHILDREN. Clinical Practice Guideline for Screening and Management of High Blood Pressure in Children and Adolescents. Pediatrics. 2017 Sep;140(3):e20171904. doi: 10.1542/peds.2017-1904. Epub 2017 Aug 21. PMID 28827377